CLINICAL TRIAL: NCT06894446
Title: Prospective, Multicenter, Open-label, Randomized (1:1 Ratio), Controlled, Parallel Study Comparing Baxter Numeta G13%E to Compounded Parenteral Nutrition (cPN) Solution to Evaluate the Efficacy and Safety of Numeta G13%E in Preterm Neonates
Brief Title: Efficacy and Safety of Numeta G13%E Compared to Compounded Parenteral Nutrition in Preterm Neonates
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision due to practice in China
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BXU512338
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Malnutrition, Infant; Enteral Feeding Intolerance
Keywords: parenteral nutrition
MeSH Terms: conditions — Infant Nutrition Disorders; Hyperphagia | interventions — Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Numeta G13%E (Experimental): Required PN intake will be determined daily based on clinical condition, calculated nutritional need and enteral nutrition (EN) intake by the attending physician in conjunction with the Investigator. Patients will receive Numeta G13%E until standard of care (SOC) discontinuation of PN, as decided by the attending physician in conjunction with the Investigator for the best interest of the patient or for a maximum of 28 days.
  Interventions: Dietary Supplement: Numeta G13%E
- Compounded Parenteral Nutrition (cPN) solution (Active Comparator): Required PN intake will be determined daily based on clinical condition, calculated nutritional need and enteral nutrition (EN) intake by the attending physician in conjunction with the Investigator. Patients will receive cPN until standard of care (SOC) discontinuation of PN, as decided by the attending physician in conjunction with the Investigator for the best interest of the patient or for a maximum of 28 days.
  Interventions: Dietary Supplement: Compounded Parenteral Nutrition (cPN) solution

INTERVENTIONS:
Dietary Supplement: Numeta G13%E — Dose selected and dosing schedule are as deemed appropriate by the ordering attending physician in conjunction with the Investigator.
  Arms: Numeta G13%E
Dietary Supplement: Compounded Parenteral Nutrition (cPN) solution — Will be administered as institutional SOC procedure for the hospital.
  Arms: Compounded Parenteral Nutrition (cPN) solution

SUMMARY:
Preterm (PT, born before 37 weeks of gestation) birth complications are the leading causes of death among children aged under 5 years globally, with nearly one million infant deaths reported in 2013. Preterm infants are born with limited nutrient stores, while birth occurs when the nutritional requirements are the highest in human life. Due to the immaturity of their gastrointestinal system, parenteral nutrition (PN) is usually required during the first weeks of life, especially in very low birth weight (VLBW) infants. Despite the availability of national and international guidelines, the initiation of PN is frequently not compliant with current recommendations, especially during the first days of life. In China, like in many other parts of the world, insufficient nutritional supply during hospital stay plays an important role in the postnatal growth restriction (PNGR) of PT infants. Several authors have recently shown that the use of standardized PN formulations can enable optimal early PN intake and can support improved growth rate without adverse consequences in PT infants. Guidelines recommend that standard PN solutions should generally be used over individualized PN solutions in the majority of pediatric and newborn patients, including VLBW infants. They also recommended that individually tailored PN solution should generally be used when the nutritional requirements cannot be met by the available range of standard PN formulations. Given the challenges of optimizing PN practice in PT infants, the aim of this study is to demonstrate non-inferiority of Numeta G13%E to classic compounding practice used for Chinese PT neonates. Please note: Secondary safety endpoints that include Adverse Events (AE) and abnormal blood results will be captured in AE section.

ELIGIBILITY:
Inclusion Criteria:

* PT birth (>28 and < 37 weeks of gestation)
* Postnatal age < 48 hours
* Medical determination of PN requirement made by the attending physician in conjunction with the Investigator
* An anticipated PN duration after inclusion of at least 5 days
* Requirement for ≥ 80 % of energy intake from PN at inclusion (PN initiation)
* Written ICF signed by the patient's legal representative

Exclusion Criteria:

* Neonates born < 28 and ≥ 37 weeks of gestation
* Neonates with a life expectancy <1 week, which means with very severe critical illness implying foreseeable intercurrent events that could jeopardize the subject's primary outcome assessment including neonates with severe septic shock;
* Neonates requiring or anticipated to undergo extracorporeal membrane oxygenation treatment;
* Neonates with inborn error of metabolism including congenital abnormality of the amino acid metabolism or a family history of such disease;
* Neonates with hyperkalemia > 5.5 mmol/L at inclusion
* Neonates with known severe pathologically elevated plasma concentrations of electrolyte at inclusion including hyperchloridemia > 120 mmol/L;
* Neonates with known severe hyperglycemia >13.9 mmol/L (250 mg/dL) at inclusion;
* Neonates with demonstrated severe hyperlipidemia or severe disorders of lipid metabolism characterized by hypertriglyceridemia > 4.5 mmol/L (400 mg/dL) at inclusion;
* Neonates with known severe liver failure including plasma ALT (GPT) concentration > 2 times the upper reference limit or conjugated (direct) bilirubin > 34 µmol/L (> 2 mg/dL) at inclusion;
* Neonates with anuria and known severe renal disorder including plasma creatinine concentration > 2 times the upper reference limit at inclusion;
* Neonates with bleeding and severe coagulation disorders including platelet count < 20×109/L at inclusion;
* Neonates with general contraindications to infusion therapy: acute pulmonary edema, overhydration;
* Neonates with known allergy to egg, soy bean or peanut proteins or to any of their active ingredients or excipients;
* Neonates undergoing concomitant treatment with ceftriaxone, even if separate infusion lines are used;
* Neonates undergoing participation in another investigational clinical study at study enrollment.

Ages: 0 Hours to 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-08-20 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Weight (SDS or z-score) at Day 14 | Baseline (first 24 hours of life) and Day 14
  The change in weight standard deviation score (SDS or z-score) from birth to 14 days of life, calculated according to reference growth chart developed to assess the growth of preterm infants. To be included in the primary endpoint analysis, patients must minimally receive PN up to Day 5.

SECONDARY OUTCOMES:
Daily Protein Intake (g/kg/day) | Day 1 to 7
  Nutritional intake from PN will be calculated as per any intravenous nutritional intake (Numeta G13%E, cPN and other sources). Nutritional intake from EN (Enteral Nutrition) will be calculated as per label for infant formula and human milk fortifier (HMF). (Protein = amino acids)
Daily Energy Intake (kcal/kg/day) | Day 1 to 7
  Nutritional intake from PN will be calculated as per any intravenous nutritional intake (Numeta G13%E, cPN and other sources). Nutritional intake from EN (Enteral Nutrition) will be calculated as per label for infant formula and human milk fortifier (HMF). Energy includes total calories, non-protein calories, glucose calories, lipid calories.
Weekly Protein Intake (g/kg/week) | Week 1, Week 2, Week 3, Week 4
  Nutritional intake from PN will be calculated as per any intravenous nutritional intake (Numeta G13%E, cPN and other sources). Nutritional intake from EN (Enteral Nutrition) will be calculated as per label for infant formula and human milk fortifier (HMF). (Protein = amino acids).
Weekly Energy Intake (kcal/kg/week) | Week 1, Week 2, Week 3, Week 4
  Nutritional intake from PN will be calculated as per any intravenous nutritional intake (Numeta G13%E, cPN and other sources). Nutritional intake from EN (Enteral Nutrition) will be calculated as per label for infant formula and human milk fortifier (HMF). Energy includes total calories, non-protein calories, glucose calories, lipid calories.
Age (hours) when minimal weight is documented | Day 1
  Measurement=hours.
Maximum weight loss (%) from birth weight | Day 1 to Day 14
  Measurement=percentage (%).
Time (hours) to regain birth weight | Day 1 to Day 14
  Postnatal age (hours) when body weight is first documented above BW after maximal weight loss.
Weight gain velocity up to Day 14 | Day 1 to Day 14
  Calculated by taking the difference between the weight at the end of treatment and the minimum weight recorded and dividing it by the total number of treatment days.
Change from Baseline in Weight (SDS or z-score) at Day 7, 14, 21 and 28 | Baseline, Day 7, Day 14, Day 21, Day 28
  Standard deviation score (SDS or z-score).
Change from Baseline in Length (SDS or z-score) at Day 7, 14, 21 and 28 | Baseline, Day 7, Day 14, Day 21, Day 28
  Standard deviation score (SDS or z-score).
Change from Baseline in Head Circumference (SDS or z-score) at Day 7, 14, 21 and 28 | Baseline, Day 7, Day 14, Day 21, Day 28
  Standard deviation score (SDS or z-score).
Weekly gain in Weight (g/kg/day) at Day 7, 14, 21 and 28 | Day 7, Day 14, Day 21, Day 28
  Measurement=g/kg/day.
Weekly gain in Length (cm/week) at Day 7, 14, 21 and 28 | Day 7, Day 14, Day 21, Day 28
  Measurement=cm/week.
Weekly gain in Head Circumference (cm/week) at Day 7, 14, 21 and 28 | Day 7, Day 14, Day 21, Day 28
  Measurement=cm/week.
Change from Baseline in Weight (SDS or z-score) at End of study | Baseline up to Week 40
  Measurement=Standard deviation score (SDS or z-score). End of Study=discharge or maximum 40 weeks post-menstrual age.
Change from Baseline in Length (SDS or z-score) at End of study | Baseline up to Week 40
  Measurement=Standard deviation score (SDS or z-score).
Change from Baseline in Head Circumference (SDS or z-score) at End of study | Baseline up to Week 40
  Measurement=Standard deviation score (SDS or z-score).
Gain in Weight (g/kg/week) from Baseline to End of study | Baseline up to Week 40
  Measurement=g/kg/week
Gain in Length (cm/week) from Baseline to End of study | Baseline up to Week 40
  Measurement=cm/week.
Gain in Head Circumference (cm/week) from Baseline to End of study | Baseline up to Week 40
  Measurement=cm/week.
Number of Clinical Characteristics by Type | Week 1 up to Week 40
  Including in-hospital deaths, necrotizing enterocolitis (NEC), late onset sepsis (LOS), bronchopulmonary dysplasia (BPD), intraventricular hemorrhage (IVH), periventricular leukomalacia (PVL), retinopathy of prematurity (ROP), and cholestasis
Duration of Clinical Characteristics by Type | Week 1 up to Week 40
  Including mechanical ventilation duration, PN duration, antibiotic duration, and in-hospital length of stay (LoS)
Adverse Events of special interest (AESIs) | Week 1 up to Week 40